CLINICAL TRIAL: NCT05430763
Title: Motor Deficits and Signal Conduction in Individuals With Williams Syndrome
Status: Withdrawn | Type: Observational
Why Stopped: No participents enrolled
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Other Study IDs: 5859-19-SMC
Record Dates: First submitted 2022-06-15; First posted 2022-06-24 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2022-06

CONDITIONS: Williams Syndrome
Keywords: Williams syndrome; Nerve conduction; Motor deficits
MeSH Terms: conditions — Williams Syndrome; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Williams syndrome: Nerve conduction test (NCT) Nerve ultrasound Clinical evaluation GAITRite walkway Motor questionnaire
- Control, age matched: Nerve conduction test (NCT) Nerve ultrasound Clinical evaluation GAITRite walkway Motor questionnaire

SUMMARY:
The current study aims to validate basic research findings of abnormal conductivity and motor abilities from a mouse model in humans. The study will measure nerve conduction properties in WS individuals and characterize motor symptoms in individuals with WS.

DETAILED DESCRIPTION:
50 individuals with WS will take part in the study. All participants will be recruited from the Williams Syndrome Clinic at Edmond and Lili Safra Children's Hospital, Sheba Medical Center directed by Prof. Doron Gothelf, MD, that coordinates treatment and research of WS in Israel. 20 control age-matched subjects will be recruited as well. A Motor Questionnaire, designed especially for this study will be filled by parents. It includes questions about gross motor, fine motor, gait and coordination characteristics of the children (Bellugi, Bihrle et al. 1990, Wilson, Kaplan et al. 2000, Wilson, Crawford et al. 2009) (General references regarding motor abilities and health).

In addition, participants will undergo the following assessments at the neuromuscular clinic and at the movement laboratory, Sheba Medical Center in collaboration with Dr. Amir Dori, Dr. Uri Givon and Dr. Meir Plotnik: (1) nerve conduction study (2) nerve ultrasound (3) neurological assessments (4) GAITRite walkway for gait analysis (5) 3-D motion analysis.

ELIGIBILITY:
Inclusion Criteria:

* WS patients.

Exclusion Criteria:

* WS patients suffering from additional neurological condition (such as epilepsy).
* Participants who will have difficulties preforming the tests may ask to be excluded.

Ages: 3 Years to 30 Years | Sex: All
Age Groups: Child, Adult
Study Population: Williams syndrome (WS) is a neurodevelopmental genetic disorder caused by a hemizygous deletion of approximately 25 genes on the long arm of chromosome 7 (7q11.23), with a prevalence of around 1 in 20,000 individuals. Individuals with WS exhibit unique social phenotype marked by strong social appetite and disinhibited social behavior. In addition, WS individuals exhibit cognitive impairments, motor deficits which are poorly defined, and several more physical and psychological phenotypes.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Nerve conduction test - Amplitude | 30 days
  This test's amplitude outcome present a nerve conduction property that can indicate aberrations in signal conduction.
Nerve conduction test - Latency | 30 days
  This test's latency outcome present a nerve conduction property that can indicate aberrations in signal conduction.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

REFERENCES:
- [Background] Barak B, Zhang Z, Liu Y, Nir A, Trangle SS, Ennis M, Levandowski KM, Wang D, Quast K, Boulting GL, Li Y, Bayarsaihan D, He Z, Feng G. Neuronal deletion of Gtf2i, associated with Williams syndrome, causes behavioral and myelin alterations rescuable by a remyelinating drug. Nat Neurosci. 2019 May;22(5):700-708. doi: 10.1038/s41593-019-0380-9. Epub 2019 Apr 22. PMID 31011227